CLINICAL TRIAL: NCT02624687
Title: Reducing Sedentary Behavior to Decrease Low Back Pain: Stand Back Study
Acronym: StandBack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Bethany Barone Gibbs, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO15060576
Record Dates: First submitted 2015-10-13; First posted 2015-12-08 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): These subjects will participate in a behavioral intervention that will focus on reducing sedentary behavior and improving self-management of pain. This will include an initial, in-person behavioral intervention and then monthly follow-up calls. In addition, subjects will receive a sit-stand desk attachment and a wrist-worn activity prompter to aid in sedentary behavior reduction.
  Interventions: Behavioral: Intervention
- Control (Placebo Comparator): These subjects will receive no intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Intervention — Participants participated in monthly, individual counselling with a trained interventionist to decrease sedentary behavior and improve pain self-management. Participants were provided with a sit-stand desk attachment and a wrist worn activity prompter..
  Arms: Intervention
Other: No intervention — No contact control
  Arms: Control

SUMMARY:
This study will test the effects of a sedentary behavior intervention on low back pain in working adults. The behavioral intervention will include the use of a sit-stand desk and a wrist-worn activity prompter that will notify participants when they have been sedentary for too long.

DETAILED DESCRIPTION:
Low back pain (LBP) is prevalent, debilitating and costly. Though exercise is a recommended treatment for LBP, outcomes are variable and adherence is often poor due to barriers such as time, sedentary jobs, and fear-avoidance of movement. Thus, the management of LBP must include a biobehavioral lifestyle treatment approach. Preliminary evidence suggests that prolonged sitting at work can exacerbate LBP, LBP is relieved shortly after prolonged sitting ends, and standing more at work can relieve pain. Thus, this proposal will examine an innovative intervention to decrease pain in patients with chronic LBP (cLBP) through a reduction in sedentary behavior. The target population will be University of Pittsburgh (UPitt) employees with cLBP who are inactive and sit at their desk for ≥20 hours/week. Over 6 months, individuals will be provided with a workstation that allows for standing while performing work duties, a wrist-worn activity device that vibrates after prolonged sedentariness, and a behavioral intervention including an initial orientation and monthly follow-up telephone contacts. This is a novel pain reduction approach that is easily incorporated into the workplace and targets a timeframe during which prolonged sitting is common. A unique aspect of the approach is that individuals with cLBP who avoid movement due to pain may especially benefit from this emerging strategy of more frequent, lifestyle activity facilitated by newly-available devices. The investigators hypothesize that this intervention will reduce pain intensity thereby leading to increased work productivity, decreased healthcare utilization, improved health-related quality of life, and improved physical function in LBP sufferers. If effective, this scalable intervention could be implemented broadly to enhance employee health.

ELIGIBILITY:
Inclusion Criteria:

1. Have chronic low back pain defined as a back pain problem that has persisted at least 3 months and has resulted in pain on at least half the days in the past 6 months
2. Oswestry low back pain index >20% to ensure a moderate level of disability is present, thus minimizing a potential floor effect
3. Currently perform deskwork at least 20 hours per week at a desk compatible with the sit-stand attachment
4. Stable employment (at least 3 months at current job and plan to stay at current job for the next 6 months)
5. Ability to obtain approval to install sit-stand workstation (i.e., from supervisor)
6. Access to internet connection and email to complete assessment surveys

Exclusion Criteria:

1. Unable to provide informed consent
2. Cardiovascular event in the last 6 months (e.g. heart attack, stoke, heart failure, revascularization procedure)
3. Presence of a comorbid condition that would limit ability to reduce sedentary behavior (e.g. currently undergoing treatment for cancer)
4. Back surgery in the past 3 months or planned in the next year
5. Presence of a medical "red flag" for a serious spinal condition (cancer, compression fracture, signs or symptoms of root compression, infection)
6. Inability to tolerate standing for any reason
7. Currently using a sit-stand desk, standing desk, or wearable activity monitor
8. Currently pregnant or planned pregnancy in the next 6 months
9. Blood pressure >159/100 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Physical Activity and Weight Management Research Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Barone Gibbs B, Hergenroeder AL, Perdomo SJ, Kowalsky RJ, Delitto A, Jakicic JM. Reducing sedentary behaviour to decrease chronic low back pain: the stand back randomised trial. Occup Environ Med. 2018 May;75(5):321-327. doi: 10.1136/oemed-2017-104732. Epub 2018 Jan 12. PMID 29330230

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: These subjects will participate in a behavioral intervention that will focus on reducing sedentary behavior and improving self-management of pain. This will include an initial, in-person behavioral intervention and then monthly follow-up calls. In addition, subjects will receive a sit-stand desk attachment and a wrist-worn activity prompter to aid in sedentary behavior reduction.
  Decreasing Sedentary Behavior
- Control: These subjects will receive no intervention.
  No intervention
Period: Overall Study
Arm/Group | Intervention | Control
Started | 13 | 14
Completed | 12 | 12
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — medical leave from work | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (9) | 51 (13) | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27
Oswestry Disability Index, % [Mean (Standard Deviation); unit: %] — The Oswestry Disability Index is measured as a percent, ranges from 1-100, with a higher score indicating worse low back pain disability.
  % | 23.6 (10.9) | 24.6 (10.3) | 24.1 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Low Back Pain Disability
Description: Oswestry Disability Index. This measurements is reported as a % (range 1-100%) where a higher score indicates worse low back pain disability.
Time Frame: 6 months
Population: ITT LOCF
Measure: Least Squares Mean (Standard Error); unit: Oswestry Disability %
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 14
Oswestry Disability % | 12.1 (2.3) | 19.6 (2.2)

2. Primary Outcome: Usual Low Back Pain
Description: Pain rated by Visual Analog Scale (Usual Back Pain). This score ranges from 1-10 where a higher score indicates worse pain.
Time Frame: 6 months
Population: ITT LOCF
Measure: Least Squares Mean (Standard Error); unit: points (out of 10)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 14
points (out of 10) | 2.87 (0.33) | 3.02 (0.32)

3. Secondary Outcome: Quality of Life (Self-reported)
Description: 36-item Short Form Survey (SF-36). This validated survey collects information on quality of life, with scores ranging from 0-100, and where higher scores indicate higher quality of life.The General Health Score is reported.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 12
points | 73.33 (11.55) | 62.08 (21.05)

4. Secondary Outcome: Mood
Description: Profile of Mood States Questionnaire. Total mood disturbance score reported here. Higher scores indicate higher mood disturbance (range 0-200 points).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 12
points | 87.25 (11.76) | 102.67 (31.58)

5. Secondary Outcome: 50-ft Walk Test
Description: Time to complete 50 ft. walk test (seconds) at usual pace. Lower time indicates better function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 12
seconds | 10.67 (1.38) | 11.09 (2.31)

6. Secondary Outcome: Chair Stand Test
Description: Time to complete 5 sit-to-stand transitions (seconds). Lower time indicates better function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 12
seconds | 10.05 (1.96) | 10.42 (2.69)

7. Secondary Outcome: Timed up and go Test
Description: Timed up and go test (seconds). A lower time indicates better function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 12
seconds | 7.49 (1.11) | 8.20 (1.43)

8. Secondary Outcome: Unloaded Reach Test
Description: Distance on an unloaded reach test (cm). Greater distance indicates better function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 12
cm | 36.2 (7.5) | 34.0 (4.9)

9. Secondary Outcome: Presenteeism
Description: Stanford Presenteeism Scale. A higher score indicates higher presenteeism (range 6-30 points).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 12
points | 27.83 (3.49) | 25.08 (5.78)

10. Secondary Outcome: Work Productivity
Description: Health and Work Questionnaire. Higher total score indicates better work productivity (range 0-240 points).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 12
points | 6.57 (0.72) | 6.61 (0.88)

11. Secondary Outcome: Physical Activity
Description: Minutes per week of moderate-to-vigorous physical activity by self-report
Time Frame: 6 months
Population: ITT LOCF
Measure: Least Squares Mean (Standard Error); unit: minutes/week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 14
minutes/week | 300 (53) | 195 (52)

12. Secondary Outcome: Sedentary Behavior
Description: Self-reported hours per day
Time Frame: 6 months
Population: ITT LOCF
Measure: Least Squares Mean (Standard Error); unit: hours/day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 14
hours/day | 7.3 (0.4) | 9.0 (0.4)

ADVERSE EVENTS:
Time Frame: Monthly during the 6 month study
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 1/13 | 5/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=13) | Control (N=14)
Worsening of Low Back Pain by >50% (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
New weakness, numbness, tingling in lower legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Medical procedure (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Outpatient correction of previous knee surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No